CLINICAL TRIAL: NCT06451744
Title: Evaluation of the Clinical Specificity of Cellular and Molecular Biomarkers Identified in Patients With Lichen Planus
Brief Title: Cellular and Molecular Biomarkers in Patients With Lichen Planus
Acronym: HELP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-048
Record Dates: First submitted 2023-07-06; First posted 2024-06-11 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Lichen Planus
MeSH Terms: conditions — Lichen Planus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Oral lichen planus erosive (Experimental): Human biological samples :
  * blood samples collection at visit 1 and 2 (6 month after first visit)
  * brushing on skin or mucous membrane lesions at visit 1
  * skin or mucous membrane biopsy at visit 1 and 2
  Interventions: Other: Blood samples collection; Other: Skin or mucous membrane brushing; Other: Skin or mucous membrane biopsy
- mucosal pemphigoid with oral lesions (Experimental): Human biological samples :
  * blood samples collection at visit 1
  * brushing on skin or mucous membrane lesions at visit 1
  Interventions: Other: Blood samples collection; Other: Skin or mucous membrane brushing
- lichen planus with scalp involvement (Experimental): Human biological samples :
  * blood samples collection at visit 1
  * brushing on skin or mucous membrane lesions at visit 1
  Interventions: Other: Blood samples collection; Other: Skin or mucous membrane brushing
- Pseudopelade of Brocq (Experimental): Human biological samples :
  * blood samples collection at visit 1
  * brushing on skin or mucous membrane lesions at visit 1
  * skin or mucous membrane biopsy at visit 1
  Interventions: Other: Blood samples collection; Other: Skin or mucous membrane brushing; Other: Skin or mucous membrane biopsy
- lichen planus with nail involvement (Experimental): Human biological samples :
  * blood samples collection at visit 1
  * brushing on skin or mucous membrane lesions at visit 1
  Interventions: Other: Blood samples collection; Other: Skin or mucous membrane brushing
- psoriasis and specific nail involvement (Experimental): Human biological samples :
  * blood samples collection at visit 1
  * brushing on skin or mucous membrane lesions at visit 1
  Interventions: Other: Blood samples collection; Other: Skin or mucous membrane brushing
- Lichenoid graft-versus-host disease (Experimental): Human biological samples :
  * blood samples collection at visit 1
  * brushing on skin or mucous membrane lesions at visit 1
  Interventions: Other: Blood samples collection; Other: Skin or mucous membrane brushing

INTERVENTIONS:
Other: Blood samples collection — 50 mL blood sample
Other: Skin or mucous membrane brushing — brushing on skin or mucous membrane lesions
Other: Skin or mucous membrane biopsy — 6 mm biopsy
  Arms: Oral lichen planus erosive; Pseudopelade of Brocq

SUMMARY:
Lichen planus (LP) is a chronic inflammatory disease of unknown aetiology, affecting the skin and mucous membranes, characterised by a CD8+ cytotoxic T-cell infiltrate, associated with epithelial cell death and disruption of the basement membrane zone. In previous work, T cell antigen receptor (TCR) repertoire studies were performed. In all patients tested, whether with erosive or non-erosive LP, unique nucleotide sequences, called clonotypes, have been identified. They appear during the process of TCR gene rearrangement. These clonotypes are specific for human papillomavirus (HPV) in blood and lesions, suggesting antigenic stimulation of these clonotypes by a viral epitope of HPV, which crosses with an epitope on keratinocytes. The diagnosis of LP is made on the basis of clinical and histological criteria, but in some patients and in some anatomical locations, the diagnosis is difficult to make and LP may be confused with other skin conditions.

DETAILED DESCRIPTION:
Lichen planus (LP) is a chronic inflammatory disease of unknown aetiology, affecting the skin and mucous membranes, characterised by a CD8+ cytotoxic T-cell infiltrate, associated with epithelial cell death and disruption of the basement membrane zone. Several triggers have been proposed for LP, including viral antigens. In previous work, T cell antigen receptor (TCR) repertoire studies were performed, i.e. investigating the diversity of TCRs expressed on the surface of an individual's lymphocyte population. In all patients tested, whether with erosive or non-erosive LP, unique nucleotide sequences, called clonotypes, have been identified. They appear during the process of TCR gene rearrangement. These clonotypes are specific for human papillomavirus (HPV) in blood and lesions, suggesting antigenic stimulation of these clonotypes by a viral epitope of HPV, which crosses with an epitope on keratinocytes. The diagnosis of LP is made on the basis of clinical and histological criteria, but in some patients and in some anatomical locations, the diagnosis is difficult to make and LP may be confused with other skin conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subject coming at the time of diagnosis of the disease before any systemic treatment, or at the time of a progressive episode of the disease, without systemic treatment or after cessation of immunomodulatory or immunosuppressive treatment
* Ability to give their consent in writing
* Must understand spoken and written French
* Affiliated to the French social security or assimilated regimes

Exclusion Criteria:

* Dermatosis exclusively localised in the skin folds or on the face (risk of scarring from biopsies)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Identification of TCR repertoire by flow cytometry | 3 years
  Determination by flow cytometry and PCR testing for TCR repertoire bias

SECONDARY OUTCOMES:
Identification of characteristic biomarkers of lichen | 3 years
  Identify complementary biomarkers characterising lichen by quantitative PCR
Identification of T CD8 clonotypes | 3 years
  Measurement of the antigenic specificity of identified T CD8 clonotypes by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Manuelle Vigiuer, Principal Investigator — CHU Reims Service de Dermatologie Avenue du Général Koenig 51092 Reims
Locations (6):
- France (6):
  - CHU de Besançon, Besançon
  - CHU Paris Seine-Saint-Denis- Hôpital Avicenne, Bobigny
  - Centre Medical de l'Institut Pasteur, Paris
  - Hôpital Saint-Louis, Paris
  - Hôpital Robert Debré, CHU de Reims, Reims
  - CHU de Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No